CLINICAL TRIAL: NCT05604976
Title: To Investigate Whether Single Catheter Primary PCI Method Can Reduce the Time Required for Primary PCI in Cases of ST Elevation Myocardial Infarction.
Brief Title: Single Catheter Primary Percutaneous Coronary Intervention Method in Patients With ST Elevation Myocardial Infarction
Acronym: SPEEDYPCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tokai University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Sho Torii, Associate Professor, Department of Cardiology, Tokai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPEEDY PCI
Record Dates: First submitted 2022-10-09; First posted 2022-11-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Primary percutaneous coronary intervention; Door-to-balloon time; guiding catheter
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Study participants are randomly divided into two groups: one in which Primary PCI is initiated with a universal guiding catheter and the other with a diagnostic catheter. Compare time from sheath insertion to first device activation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SC-PCI (Experimental): Primary PCI is initiated with a universal guiding catheter (Ikari left). The guiding catheter is used to contrast the left and right coronary arteries and PCI is started directly. This method does not require a catheter exchange. It is Single Catheter PCI (SC-PCI) method.
  Interventions: Device: Percutaneous coronary intervention
- Conventional (Active Comparator): Primary PCI is initiated with a diagnostic catheter. The catheter is used to contrast one of the coronary arteries. Then, the catheter is replaced with a contralateral side diagnostic catheter. Then, the catheter is replaced with a guiding catheter and PCI is started.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Primary PCI for ST elevation myocardial infarction initiating with a universal guiding catheter or an angiographic catheter

SUMMARY:
The goal of this clinical trial is to test reducing procedure time of percutaneous coronary intervention (PCI) in ST elevation myocardial infarction by single catheter PCI (SC-PCI) method. The main question it aims to answer is:

• [question 1] SC-PCI method is skipping catheter exchange with use of a right and left dual purpose universal guiding catheter Ikari Left curve. Does SC-PCI method reduce PCI procedure time? Participants will be randomly assigned to SC-PCI method or conventional method and emergency PCI is performed.

Researchers will compare time from sheath insertion to first device activation between the SC-PCI method and the conventional method.

DETAILED DESCRIPTION:
<<Background>>

Acute ST-segment elevation myocardial infarction is a disease of high acute-phase mortality rate, but the life can be saved by implementing emergency percutaneous coronary intervention (PCI). Its efficacy is higher than that of thrombolytic therapy. Moreover, shortening of total ischemia time reduces the mortality rate and can promote recovery of cardiac function. The total ischemia time can be classified into the time from onset to arrival at hospital and the time from arrival at hospital to recanalization of coronary artery (Door-to-balloon time), and shortening of time in all steps is recommended. Various methods, including the part of transportation to hospital and from arrival at hospital to treatment room, are proposed, but there is no effective method for shortening of procedure time for PCI.

Since the right and left dual-purpose universal guiding catheter can be inserted into both the left and right coronary arteries, the time for replacement of catheter can be shortened. Since IKARI Curve catheter is considered to be the most excellent catheter as the universal guiding catheter, it is considered useful for shortening of reperfusion time in myocardial infarction.

<<Objectives.>>

There are a lot of reports that decreased mortality and improvement of cardiac function are observed by shortening of the time from onset of acute myocardial infarction to recanalization. However, shortening of catheterization time, a part of the time, has not been examined. In 60 patients in a single-center retrospective study performed in Tokai University, the time from arterial puncture to reperfusion was shortened, and the time from arrival at hospital to reperfusion was also shortened. In 1275 patients in a multi-center retrospective study, moreover, the time from arterial puncture to reperfusion was significantly shortened by 4 minutes, and a significant decrease was also observed in the time from arrival at hospital to reperfusion. The Door-to-balloon time at this time was 68±46 minutes in the SC-PCI group and 76±51 minutes by the conventional method. Moreover, the time from insertion of sheath to balloon was 19±14 minutes in the SC-PCI group and 23±14 minutes by the conventional method. In addition, shortening of fluoroscopy time was also observed.

Based on this result, the information shall be collected from prospective multi-center randomized study and analyzed to verify that the right and left dual-purpose guiding catheter is useful for shortening of reperfusion time in myocardial infarction.

<<Methods.>>

Multi-center cooperative prospective interventional study, 2-group comparative study, and randomization <Conventional method> If the patients are allocated to this group, the procedure shall be started with an angiographic catheter.

An angiographic catheter is a catheter classified into a special treatment material, "Angiographic Catheter (General Model) Request Code 738180000," and approved for insurance coverage. The catheters adopted by each institution shall be used.

Coronary angiography shall be performed using an angiographic catheter, and PCI shall be performed by replacing to a guiding catheter. There are methods in which a catheter for angiography on right and left sides is performed, a dual-purpose contrast catheter is used, and one contrast catheter and guiding catheter are used, but any method is acceptable if the procedure is started from an angiographic catheter.

<SC-PCI method> When allocated to this group, the procedure shall be started with a guiding catheter of Ikari L Curve. As the Ikari L Curves approved for insurance coverage in Japan, 52 types exist by catalogue according to the difference in diameter and form, of 6 shafts of 5 companies (attached documents). Any of them shall be used. Thereafter, the right and left coronary angiography shall be performed with one right and left dual-purpose guiding catheter, and then PCI shall be performed.

Even if allocated to any group, Synergy stent shall be used when a stent is placed in coronary artery dilation.

A prospective randomization study shall be performed to reduce the bias. For the Sheath-to-First device activation time, a primary endpoint, a test of superiority shall be performed. For the Door-to-balloon time, a secondary endpoint, a test of non-inferiority shall be performed, and if the non-inferiority is demonstrated, a test of superiority shall also be performed.

The primary endpoint shall be analyzed by Intention-to-treat. The operators who can participate in this study shall take charge of any group, and who are the PCI operators who have used the Ikari L Curve guiding catheter on the right coronary artery in at least 5 patients and left coronary artery in at least 5 patients.

<<Number of Target Patients and Rationales for Setting>>

<Number of target patients> 400 patients in total (200 patients for SC-PCI method, 200 patients for conventional method) <Rationale for setting> In a multicenter retrospective study, the time from insertion of sheath to balloon (S2B) was 19±14 minutes in the SC-PCI group and 23±14 minutes for the conventional method. When testing at the level of significance of 0.05 and the power of 0.8 based on this value, the number of patients will become 388. Considering 3% dropout cases, registration of a total of 400 patients is planned.

A secondary endpoint, the D2B time was 68±46 minutes in the SC-PCI group and 76±51 minutes for the conventional method as a result of retrospective study. When testing at the level of significance of 0.05 and the power of 0.8 based on this value, the number of patients will become 1160. Therefore, the power is insufficient to show significance in the analysis of D2B time, and a non-inferiority test shall be performed. The margin of noninferiority is set at 1.3. If the D2B time by the conventional method is 76 minutes, the 1.3 times longer time is 98.8 minutes, and the difference is 22.8 minutes. In the treatment of myocardial infarction, the difference of 23 minutes or more is considered to be inferior from the standpoint of expert, and therefore it was set. Non-inferiority test shall be performed based on the 95% confidence interval (test of two-sided 5% or one-sided 2.5%) of the difference from mean value. If non-inferiority is shown, the test of superiority shall also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 21 years or older
2. Acute ST-segment elevation myocardial infarction
3. Patients indicated for Primary PCI within 12 hours after onset

Exclusion Criteria:

1. Patients with shock requiring insertion of Impella, ECMO or IABP before PCI
2. Patients requiring cardiopulmonary resuscitation due to cardiac arrest
3. Patients requiring temporary pacemaker due to bradycardia
4. Patients undergoing dialysis
5. Patients judged by the attending physician to be inappropriate for registration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Sheath-to-first device activation time | the end of PCI
  Time from insertion of sheath to reperfusion treatment apparatus (First device activation)

SECONDARY OUTCOMES:
Door-to-balloon time | the end of PCI
  Time from arrival at hospital to reperfusion treatment apparatus (First device activation)
Total ischemia time | the end of PCI
  Time from the onset of myocardial infarction to achievement of TIMI 3 reperfusion
Fluoroscopy time and fluoroscopy dose | the end of PCI
  Radiation dose assessed as fluoroscopy time and dose
Amount of contrast medium | the end of PCI
  Dose of contrast medium used during PCI procedure
Number of catheters used | the end of PCI
  Total number of catheters used during the PCI procedure
Hospital expense | 30 days
  Total cost required for the total hospital stay
All-cause mortality and cardiovascular mortality at 30 days | At 30 days from the onset of STEMI
  All-cause mortality and cardiovascular mortality at 30 days
Hemorrhagic complication rate at 30 days | At 30 days from the onset of STEMI
  BARC 3 or 5 hemorrhagic complications
All-cause mortality and cardiovascular mortality at 1 year | 1 year after the randomization
  All-cause mortality and cardiovascular mortality at 1 year
Success rate of SC-PCI method | the end of PCI
  Success of SC-PCI method is defined as diagnostic angiography and PCI is performed using a single universal guiding catheter, Ikari left.

CONTACTS AND LOCATIONS:
Overall Officials: Sho Torii, MD, Principal Investigator — Tokai University
Locations (1):
- Tokai University Hospital, Isehara, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No
There are no plans to obtain IPD consent from patients.

REFERENCES:
- [Result] Lee KH, Torii S, Oguri M, Miyaji T, Kiyooka T, Ono Y, Asada K, Adachi T, Takahashi A, Ikari Y. Reduction of door-to-balloon time in patients with ST-elevation myocardial infarction by single-catheter primary percutaneous coronary intervention method. Catheter Cardiovasc Interv. 2022 Feb;99(2):314-321. doi: 10.1002/ccd.29797. Epub 2021 May 31. PMID 34057275
- [Result] Torii S, Fujii T, Murakami T, Nakazawa G, Ijichi T, Nakano M, Ohno Y, Shinozaki N, Yoshimachi F, Ikari Y. Impact of a single universal guiding catheter on door-to-balloon time in primary transradial coronary intervention for ST segment elevation myocardial infarction. Cardiovasc Interv Ther. 2017 Apr;32(2):114-119. doi: 10.1007/s12928-016-0395-z. Epub 2016 Apr 28. PMID 27125428
- [Result] Youssef AA, Hsieh YK, Cheng CI, Wu CJ. A single transradial guiding catheter for right and left coronary angiography and intervention. EuroIntervention. 2008 Jan;3(4):475-81. doi: 10.4244/eijv3i4a85. PMID 19736091
- [Result] Ikari Y, Masuda N, Matsukage T, Ogata N, Nakazawa G, Tanabe T, Morino Y. Backup force of guiding catheters for the right coronary artery in transfemoral and transradial interventions. J Invasive Cardiol. 2009 Nov;21(11):570-4. PMID 19901410
- [Result] Ikari Y, Nagaoka M, Kim JY, Morino Y, Tanabe T. The physics of guiding catheters for the left coronary artery in transfemoral and transradial interventions. J Invasive Cardiol. 2005 Dec;17(12):636-41. PMID 16327043
- [Result] Ikari Y, Nakajima H, Iijima R, Aoki J, Tanabe K, Nakayama T, Miyazawa A, Hatori M, Kyouno H, Tanimoto S, Amiya E, Nakazawa G, Onuma Y, Hara K. Initial characterization of Ikari Guide catheter for transradial coronary intervention. J Invasive Cardiol. 2004 Feb;16(2):65-8. PMID 14760193
- [Result] Ikari Y, Ochiai M, Hangaishi M, Ohno M, Taguchi J, Hara K, Isshiki T, Tamura T, Yamaguchi T. Novel guide catheter for left coronary intervention via a right upper limb approach. Cathet Cardiovasc Diagn. 1998 Jun;44(2):244-7. doi: 10.1002/(sici)1097-0304(199806)44:23.0.co;2-l. PMID 9637453
- See also: Homepage about Ikari curve — https://ikaricurve.com